CLINICAL TRIAL: NCT01157832
Title: Evaluation of the Acute Effect of Water-Pipe Smoking on the Respiratory System
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Other Study IDs: RMC-0219-09
Record Dates: First submitted 2010-07-06; First posted 2010-07-07 (Estimated); Last update posted 2013-06-11 (Estimated); Status verified 2013-06

CONDITIONS: Carboxyhemoglobin; Vital Signs; Fractional Exhaled NO; Exhaled Breath Condensate
Keywords: water pipe smoking acute effect

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Title: The acute effect of water pipe smoking on exhaled nitric oxide (eNO) and exhaled breath condensate (EBC) pulmonary function tests in healthy volunteers

Objectives: To evaluate the acute effect of one cession of water pipe smoking on airway inflammation as assessed by exhaled nitric oxide (eNO) and exhaled breath condensate (EBC) in healthy volunteers.

Design: Prospective study evaluating these parameters before and after 30 minutes of water pipe smoking . The changes in inflammatory parameters pre and post smoking will be evaluated blindly.

Sample size: 100 participants Participant selection: Adults subjects who regularly smoke water pipe . Intervention: Each subject will undergo evaluation including a respiratory questionnaire , pulmonary function tests , exhaled nitric oxide (eNO) and exhaled breath condensate (EBC) and carboxy- hemoglobin levels . All measurements will be evaluated before and after one cession of 30 minutes water pipe smoking

Primary outcome parameter: Change in carboxy- hemoglobin Secondary outcome parameter:Change in peripheral eosinophils count, pulmonary function tests, change in FeNO, and in inflammatory parameters in EBC before and after water pipe smoking

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 Y.O.
* Have smoked Water-pipe at least once before.

Exclusion Criteria:

* Breast feeding Women.
* S/P Bacterial Or Viral infection, Last 2 weeks
* P.O. Steroids
* Water-pipe smoking, last 24 hours
* Cigarette smoking, last 6 hours
* Intensive exposure to smoke (fire), last 24 hours
* S/P Intensive Care Hospitalization, last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal People who have smoked Water-pipe, at least once before.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2009-11; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
carboxy- hemoglobin | before and immediatly after 30 min of smoking
  blood test

SECONDARY OUTCOMES:
Eosinophils count | before and immediatly after 30 min of smoking
  blood test
heart rate | before and immediatly after 30 min of smoking
  heart beats count
Respiratory rate | before and immediatly after 30 min of smoking
  Respiratory rate
Blood pressure | before and immediatly after 30 min of smoking
  Non Invasive Blood pressure mesaurement
Spirometry | before and immediatly after 30 min of smoking
  Pulmonary function test
Visual Analog Score 1-10 (1=bad 10=good) | before and immediatly after 30 min of smoking
  Questionnaire
Exhaled breath Condensate | before and immediatly after 30 min of smoking
  R-tube tests
Fractional Exhaled NO | before and immediatly after 30 min of smoking
  Exhaled NO test

CONTACTS AND LOCATIONS:
Overall Officials: Lea Bentur, Prof., Principal Investigator — Rambam Health Care Campus
Locations (2):
- Israel (2):
  - RAMBAM Health Care Campus, Haifa, Israel
  - Rambam Medical Center, Haifa

REFERENCES:
- [Background] Nakkash R, Khalil J. Health warning labelling practices on narghile (shisha, hookah) waterpipe tobacco products and related accessories. Tob Control. 2010 Jun;19(3):235-9. doi: 10.1136/tc.2009.031773. PMID 20501497
- [Background] Daher N, Saleh R, Jaroudi E, Sheheitli H, Badr T, Sepetdjian E, Al Rashidi M, Saliba N, Shihadeh A. Comparison of carcinogen, carbon monoxide, and ultrafine particle emissions from narghile waterpipe and cigarette smoking: Sidestream smoke measurements and assessment of second-hand smoke emission factors. Atmos Environ (1994). 2010 Jan 1;44(1):8-14. doi: 10.1016/j.atmosenv.2009.10.004. PMID 20161525
- [Background] Eissenberg T, Shihadeh A. Waterpipe tobacco and cigarette smoking: direct comparison of toxicant exposure. Am J Prev Med. 2009 Dec;37(6):518-23. doi: 10.1016/j.amepre.2009.07.014. PMID 19944918
- [Background] Maziak W. The waterpipe: time for action. Addiction. 2008 Nov;103(11):1763-7. doi: 10.1111/j.1360-0443.2008.02327.x. Epub 2008 Sep 4. PMID 18778388
- [Result] Chaouachi K. Lessons from the recent case of CO poisoning due to shisha (hookah, narghile) tobacco smoking in Singapore. Int J Emerg Med. 2010 Feb 6;3(1):67-8. doi: 10.1007/s12245-009-0139-2. No abstract available. PMID 20414388
- [Result] Lim BL, Lim GH, Seow E. Case of carbon monoxide poisoning after smoking shisha. Int J Emerg Med. 2009 Mar 11;2(2):121-2. doi: 10.1007/s12245-009-0097-8. PMID 20157455
- [Derived] Hakim F, Hellou E, Goldbart A, Katz R, Bentur Y, Bentur L. The acute effects of water-pipe smoking on the cardiorespiratory system. Chest. 2011 Apr;139(4):775-781. doi: 10.1378/chest.10-1833. Epub 2010 Oct 28. PMID 21030492